

Prospective Clinical Evaluation of the Safety and Efficacy of NON-INVASIVE Electronic Stimulation for Improvement of Muscle Strength and Toning, Circumferential Reduction of the Core and Extremities

Sponsor: Lutronic, Inc. Funded by: Lutronic, Inc.

Date: September 8, 2021 Clinical Protocol Number: AFL19006 Version number: 2.0

# Sponsor Statement and Signature Page

Company Name: Lutronic, Inc.

Address: 19 Fortune Drive

Billerica, MA 01821

Telephone: 888-588-7644

The investigation will be conducted in compliance with the clinical investigation plan (CIP), GCP, EN ISO 14155, the Declaration of Helsinki, and regulatory authority requirements.

Lutronic, Inc. (hereinafter "Study Sponsor") maintains responsibility for the ongoing safety of this clinical trial involving the evaluation of the Genius System. Study Sponsor will promptly notify all investigators, the responsible IRB(s), and the regulatory authorities of any findings from ongoing trial monitoring activities that could adversely affect the safety of subjects, impact the conduct of the clinical study, or alter the IRB's approval to continue the study, specifically within 5 working days of making an Unanticipated Adverse Device Effect (UADE) determination or 15 working days after first receiving notice of the UADE, within 10 days for Serious Adverse Event reports, and at least annually for routine reports. In the event that participant safety could be directly affected by study results after the study has ended, Study Sponsor will notify all investigators of these results to enable investigators to consider informing participants as soon as possible or at least within one year of study closure. The following individuals are responsible for the content of the Clinical Investigational Plan:

| Paul Cardarelli | Date |
|---------------------------------------------------|------|
| Director, Clinical Research & Product Development | |

## **Contact Information**

Protocol Number: AFL19006

Sponsor: Lutronic Global

19 Fortune Dr. Billerica, MA 01821

Lutronic Contact Information: Paul Cardarelli

Director, Clinical Research & Product Development

Phone: 888-588-7644

Email: pcardarelli@lutronic-usa.com

Protocol Number: AFL19006 

Site Contact Information: Primary Investigator

Omar A. Ibrahimi, M.D., Ph.D.

19 Fortune Dr. Billerica, MA 01821

Email: omar.ibrahimi@gmail.com

Tel: (203) 428-4440 Fax: (203)890-9449

ANNE M. CHAPAS, M.D.

Union Square Laser Dermatology

19 Union Square West New York, NY 10003 Phone: (212) 366-5400 Fax: (212) 366-5461

If you have any questions or complaints about your rights as a research subject, contact:

Allendale IRB

Telephone: (860)434-5872

Fax: (860)434-5892 rta1ali1@aol.com

# Statement of Compliance

I have thoroughly read and reviewed this clinical investigation plan (CIP) and hereby agree to participate in this clinical trial sponsored by Lutronic, Inc. I agree to conduct this investigation according to the requirements of the CIP provided by the Study Sponsor and in accordance with Good Clinical Practice (GCP) as required by EN ISO 14155, the Declaration of Helsinki, Investigational Device Exemption (21 CFR Part 812), Protection of Human Subjects (45 CFR Part 46), and other applicable FDA regulations, and regulations of other relevant regulatory authorities and conditions imposed by the reviewing Institutional Review Board (IRB) or Ethics Committee (EC). I agree that no deviation from, or changes to the CIP will take place without prior agreement from the sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants. I agree to ensure that appropriate informed consent is obtained from all subjects prior to inclusion in this study. I also agree to supervise all testing of the device involving human subjects, and to report to the Study Sponsor, within 24 hours, any adverse event that is serious, whether considered treatment-related or not. I am aware that the Study Sponsor reserves the right to discontinue this investigation at any time.

I understand that this investigation will be monitored by the Study Sponsor and/or a designee contracted or employed by the Study Sponsor. This monitoring will involve periodic inspection of my investigational site and ongoing review of the data that is submitted by me to the Study Sponsor. All study data will be scanned and uploaded within 1 week after the study visit. I am also aware that I may be inspected by a representative of the relevant regulatory authorities, including the United States Food and Drug Administration, to verify compliance with applicable regulations related to clinical research on human subjects.

My current curriculum vitae and the curriculum vitae of physicians/licensed practitioners at this institution who will participate as co-investigators/sub-investigators in this study will be provided to the Study Sponsor. This curriculum vitae will include the extent and type of our relevant experience with pertinent dates and locations. All personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I certify that I have not been involved in an investigation that was terminated for non-compliance at the insistence of the Study Sponsor, the IRB or EC, or other regulatory authorities. I agree to provide the Study Sponsor sufficient, accurate financial disclosure information. I also agree to update financial disclosure information if any relevant changes occur during the investigation and for one year following the completion of the study.

I understand that this CIP and the trial results are confidential, and I agree not to disclose any such information to any person other than a representative of the Study Sponsor or the relevant competent authorities without the prior written consent of the Study Sponsor.

Accepted by:

| Principal Investigator Signature | Principal Investigator Name | Date |
|----------------------------------|-----------------------------|----------|
| Co-/Sub-Investigator Signature | Co-/Sub-Investigator Name | <br>Date |
| Co-/Sub-Investigator Signature | Co-/Sub-Investigator Name | <br> |

Protocol Number: AFL19006 

# List of Abbreviations

| TERM | DEFINITION | TERM | DEFINITION |
|---|---|---|---|
| AE | Adverse Event | ICH E6 | International Conference on<br>Harmonization Guidance for Industry,<br>Good Clinical Practice: Consolidated<br>Guidance |
| ADE | Adverse Device Effect | ICMJE | International Committee of Medical Journal Editors |
| ANCOVA | Analysis of Covariance | IDE | Investigational Device Exemption |
| BMI | Body Mass Index | IFU | Instructions for Use |
| CFR | Code of Federal Regulations | ISO | International Organization for Standardization |
| CGAIS | Clinician Global Aesthetic Improvement<br>Scale | IRB | Institutional Review Board |
| CIP | Clinical Investigation Plan | МОР | Manual of Procedures |
| CMP | Clinical Monitoring Plan | NRS | Numeric Rating Scale for pain assessment |
| CRF | Case Report Form | OHRP | Office for Human Research Protections |
| CRO | Contract Research Organization | PI | Principal Investigator |
| CV | Curriculum Vitae | PSQ | Patient Satisfaction Questionnaire |
| DCC | Data Coordination Center | QA | Quality Assurance |
| DSMB | Data Safety Monitoring Board | QC | Quality Control |
| EC | Ethics Committee | RF | Radiofrequency |
| eCRF | Electronic Case Report Form | Rhytidectomy | Mini facelift |
| ETE | Expected Treatment Effect | SAE | Serious Adverse Event |
| FDA | Food and Drug Administration | SAP | Statistical Analysis Plan |
| FDAAA | Food and Drug Administration Amendments Act of 2007 | SADE | Serious Adverse Device Effect |
| GAIS | Global Aesthetic Improvement Scale | SGAIS | Subject Global Aesthetic Improvement<br>Scale |
| GCP | Good Clinical Practice | SMC | Safety Monitoring Committee |
| GLP | Good Laboratory Practice | SOP | Standard Operating Procedure |
| GMP | Good Manufacturing Practice | UADE | Unanticipated Adverse Device Effect |
| НІРАА | Health Information Portability and Accountability Act | USA | United States of America |
| IB | Investigator's Brochure | | |
| ICH | International Committee on Harmonization | | |

Protocol Number: AFL19006 Page **5** of **35** 

# **Protocol Synopsis**

| Protocol Number: | AFL19006 |
|---|---|
| Protocol Title: | Prospective Clinical Evaluation of the Safety and Efficacy of NON-INVASIVE Electronic Stimulation for Improvement of Muscle Strength and Toning, Circumferential Reduction of the Core and Extremities |
| Investigational Devices: | The Accufit Electrical Muscle Stimulation device is an FDA cleared two-channel muscle stimulator that provides up to 8 electrodes with unique waveforms for muscle stimulation. |
| Development Phase: | Evaluation |
| Study Objective: | The objective of this clinical study is to assess the safety and efficacy of a novel electrical |
| | stimulation device for use in improving muscle strength and toning of the core and extremities. |
| Brief Study Overview: | Open-label, baseline-controlled, multi-center study evaluating an electrical muscle stimulation system for Improvement of Muscle Strength and Toning, Circumferential Reduction of the Core and Extremities The study will enroll up to 60 subjects desiring and to improve muscle strength and tone and circumferential reduction in their core and extremities. Each subject will receive up to 8 bi-weekly treatments over a 4-week period. Follow up visits planned for 30- and 90-days post treatment. Measurement outcomes will be compared to baseline. |
| Number of Sites | Up to 6 sites |
| Enrolling Participants: | |
| Sample Size: | The study will enroll up to 60 male and female subjects ≥ 18 years to 60 years of age who are seeking to improve muscle strength and tone in the extremities. |
| Subject Population: | Healthy, female and male adult subjects age 18 to 60 years who meet the inclusion/exclusion criteria. |
| Inclusion Criteria: | <ol> <li>Able to read, understand and voluntarily provide written informed consent.</li> <li>Healthy male or female, ≥ 18 years to 65 years of age seeking treatment for improved muscle strength and muscle toning in their core and extremities.</li> <li>Subject is determined to be physically fit and agrees to not making any major changes in their diet or lifestyle during the study.</li> <li>Able and willing to comply with the treatment/follow-up schedule and requirements.</li> <li>Women of child-bearing age are required to be using a reliable method of birth control at least 3 months prior to study enrollment and for the duration of the study as well as have a negative Urine Pregnancy test at baseline.</li> </ol> |
| Exclusion Criteria: | <ol> <li>Pregnant in the last 3 months, intending to become pregnant, postpartum or nursing in the last 6 months.</li> <li>Any previous liposuction/lipo-sculpture or any type of surgical procedure in the treatment area in the past 12 months.</li> <li>History of immunosuppression/immune deficiency disorders (including AIDS and HIV infection) or use of immunosuppressive medications, 6 months prior to and during the study.</li> <li>History of hyperlipidemia, diabetes mellitus, hepatitis, blood coagulopathy or excessive bleeding.</li> <li>Having a history of skin cancer or any other cancer in the areas to be treated, including presence of malignant or premalignant pigmented lesions.</li> <li>Having a permanent implant in the treatment area such as metal plates or an injected chemical substance such as silicone in the treatment area.</li> <li>Suffering from significant skin conditions in the treatment area or inflammatory skin conditions including but not limited to open lacerations, abrasions, herpes sores, cold sores, active infections.</li> <li>Poor skin quality (severe laxity).</li> <li>Abdominal wall, muscular abnormality or hernia on physical examination.</li> <li>As per the investigator's discretion, any physical or mental condition which may make it unsafe for the subject to participate.</li> </ol> |

Protocol Number: AFL19006 

| | <ol> <li>Subjects unwilling or unable to adhere to all study requirements for treatment and<br/>follow-up.</li> </ol> |
|---|---|
| | 12. Investigator may exclude any subject at any time at his/her discretion. |
| Primary Endpoint: | Photographic evaluation by an independent, blinded reviewer with correct identification of pretreatment baseline images when compared to post-treatment images taken at follow up visits. |
| Secondary Endpoints: | <ol> <li>Global Aesthetic Improvement grading by Expert Clinician.</li> <li>Improvement of muscle strength as measured by a dynamometer at follow up visits compared to baseline measurements.</li> <li>Reduction in core circumference as measured by Seca Circumferential System at follow</li> </ol> |
| | up visits compared to baseline measurement. 4. To assess subject satisfaction using Satisfaction Survey at each follow up visit. |
| Safety Endpoints: | Subject's assessment of discomfort as measured by a 0-10 numeric rating scale. Subjects experiencing a treatment-related adverse event (AE). |
| Study Duration: | The duration from when the study opens to enrollment for 12 months. |
| Participant Duration: | 7 months |

Protocol Number: AFL19006

| Table of Contents | |
|----------------------------------------------------------------------|----|
| Sponsor Statement and Signature Page | 2 |
| Contact Information | 2 |
| Statement of Compliance | 4 |
| List of Abbreviations | 5 |
| Protocol Synopsis | 6 |
| 1. KEY ROLES | 11 |
| 1.1 Internal Responsibilities | 11 |
| 2. INTRODUCTION: BACKGROUND INFORMATION AND SCIENTIFIC RATIONALE | 11 |
| 2.1 Background Information | 11 |
| 2.1.1 Device Name and Indications for Use | 11 |
| 2.1.2 Mechanism of Actions | 11 |
| 2.1.3 Device Overview | 11 |
| 2.2 Rationale | 12 |
| 2.3 Potential Risks and Benefits | 12 |
| 2.3.1 Known Potential Risks | 12 |
| 2.3.2 Contraindications | 12 |
| 2.3.3 Known Potential Benefits | 12 |
| 3. OBJECTIVES AND PURPOSE | 13 |
| 3.1 Study Objectives | 13 |
| 3.2 Study Endpoints | 13 |
| 3.2.1 Primary Endpoint | 13 |
| 3.2.2 Secondary Endpoints | 13 |
| 4. STUDY DESIGN AND ENDPOINTS | 13 |
| 4.1 Description of the Study Design | 13 |
| 4.2 Duration of Study | 13 |
| 5. SUBJECT ENROLLMENT AND WITHDRAWAL | 14 |
| 5.1 Participant Inclusion Criteria | 14 |
| 5.1.1 Informed Consent | 14 |
| 5.1.2 Pre-treatment Recruiting/Screening | 14 |
| 5.1.2.1 Screen Failures | 14 |
| 5.1.3 Inclusion Criteria | 14 |
| 5.1.4 Participant Exclusion Criteria | 15 |
| 5.2 Strategies for Recruitment and Retention | 15 |
| 5.2.1 Subject Payment | 16 |
| 5.3 Participant Withdrawal or Termination | 16 |
| 5.4 Premature Termination or Suspension of the Study or a Study Site | 16 |

| FI | ectronic | Stimulation | for Mus | cle Toning | and Circun | nferential | Reduction |
|---|---|---|---|---|---|---|---|
| | lectionic | Stilliulation | TOT IVIUS | cie ronning | and Circui | merendar | Reduction |

| 6. | STUD | Y PROCEDURES AND SCHEDULE | 16 |
|---|---|---|---|
| 6 | 5.1 | Photography | 16 |
| 6 | 5.2 | Study Schedule | 17 |
| | 6.2.1 | STUDY SPECIFIC PROCEDURES | 17 |
| 6 | 5.3 | LABORATORY EVALUATION | 17 |
| 6 | 5.4 | Screening & Baseline Assessment (Visit 1) | 17 |
| 6 | 5.5 | Study Treatment | 18 |
| | 6.5.1 | Subject Preparation for Study Treatment | 18 |
| | 6.5.2 | Study Treatment (Visits 1-12) | 18 |
| | 6.5.3 | Acute Responses | 19 |
| | 6.5.4 | Post- Care Instructions | 19 |
| | 6.5.5 | Schedule of Activities | 19 |
| | 6.5.6 | Safety Assessments | 20 |
| | 6.5.7 | Unscheduled Visit | 20 |
| 6 | 5.6 | Study Treatment | 20 |
| | 6.6.1 | Subject Preparation for Study Treatment | 20 |
| | 6.6.2 | Study Treatment | 20 |
| | 6.6.3 | Acute Responses | 20 |
| | 6.6.4 | Post- Care | 20 |
| 6 | 5.7 | Concomitant Medications | 20 |
| 7. | ASSE | SSMENT OF SAFETY | 21 |
| 7 | 7.1 | Specifications of Safety Parameters | 21 |
| | 7.1.1 | Definition of an Expected Treatment Effect (ETE) and an Adverse Event (AE) | 21 |
| | 7.1.2 | Definition of Serious Adverse Event (SAE) | 21 |
| | 7.1.3 | Definition of Unanticipated Adverse Device Effects (Events) | 21 |
| 7 | 7.2 | Classification of an Event | 22 |
| | 7.2.1 | Severity of Event | 22 |
| | 7.2.2 | Relationship to the Investigational Device | 22 |
| | 7.2.3 | Expectedness | 22 |
| 7 | 7.3 | Time Period and Frequency for Event Assessment and Follow-up | 22 |
| 7 | 7.4 | Reporting Procedures | 23 |
| | 7.4.1 | Adverse Event Reporting | 23 |
| | 7.4.2 | Serious Adverse Event Reporting | 23 |
| | 7.4.3 | Unanticipated Adverse Device Effect Reporting | 23 |
| | 7.4.4 | Reporting of Pregnancy | 23 |
| | 7.4.5 | Reporting of Deaths | 24 |
| 8. | CLINI | CAL MONITORING | 24 |

| Electronic Stimulation | on for Muscle Toning and Circumferential Reduction | Version 2.0 |
|---|---|---|
| 9. STATISTICAL AI | NALYSIS | 25 |
| 9.1 Statistica | l and Analytical Plans | 25 |
| 9.2 Analysis | Datasets | 26 |
| 9.3 DESCRIP | TION OF STATISTICAL METHODS | 26 |
| 9.4 SAFETY A | NALYSES | 26 |
| 9.6 BASELINE | DESCRIPTIVE STATISTICS | 27 |
| 9.7 Analysis | of Primary Endpoints | 27 |
| 9.8 Analysis | of Secondary Endpoints | 27 |
| 10. SOURCE DO | CUMENTS AND ACCESS TO SOURCE DATA/ DOCUMENTS | 28 |
| 11. ETHICS/PRO | TECTION OF HUMAN SUBJECTS | 28 |
| 11.1 Ethical St | andard | 28 |
| 11.2 Institutio | nal Revthighiew Board | 28 |
| 11.3 Informed | Consent Process | 29 |
| 11.3.1 Cor | sent/Assent and Other Informational Documents Provided to Participants | 29 |
| 11.3.2 Cor | sent Procedures and Documentation | 29 |
| 11.4 Participa | nt and Data Confidentiality | 29 |
| 12. DATA HAND | LING AND RECORD KEEPING | 29 |
| 12.1 Data Coll | ection and Management Responsibilities | 29 |
| 12.2 Investiga | tor Records and Reports | 30 |
| 12.2.1 Inve | estigator Records | 30 |
| 12.2.2 Inve | estigator Reports | 30 |

12.3

12.4

12.5

13.1

13.2

References

APPENDIX

13.

14.

Study Records Retention

**Publication and Data Sharing Policy** 

**Protocol Deviations** 

STUDY ADMINISTRATION

**Study Investigators** 

Amendment Policy

CONFLICT OF INTEREST POLICY

PROTOCOL REVISIONS LOG

31

31

32

32

32

32

33

34

35

## 1. KEY ROLES

Persons serving in key roles in the conduct or oversight of this clinical trial are listed in Table 1.1-1 below.

#### 1.1 Internal Responsibilities

**TABLE 1: INTERNAL RESPONSIBILITIES** 

| Name | Function | Address |
|---|---|---|
| Lutronic Aesthetics Sponsor | | 19 Fortune Drive |
| | | Billerica, MA 01821 |
| | | Phone: 888.588.7644 |
| Paul Cardarelli | Clinical Research Director | Phone: 888.588.7644<br>Email: <u>pcardarelli@lutronic-usa.com</u> |

# 2. INTRODUCTION: BACKGROUND INFORMATION AND SCIENTIFIC RATIONALE

#### 2.1 BACKGROUND INFORMATION

In 1761 Luigi Galvani provided scientific evidence that current can activate muscle. Electrical Muscle Stimulation is known to assist in muscle contraction.

#### 2.1.1 Device Name and Indications for Use

Magnet-based and Direct muscle stimulation devices are commonly used to generate current flow through the muscles in order to activate the muscle. The Accufit Electrical Muscle Stimulation device is an FDA cleared device having a two-channel stimulator that provides up to 8 electrodes with waveforms of interferential and biphasic for muscle stimulation. The Accufit system is indicated for relaxation of muscles, muscle re-education, reduction of pain and increased local blood circulation.

## 2.1.2 Mechanism of Actions

Muscle stimulation technology has been around for many decades and has been shown to be safe and effective for a variety of clinical applications. The foundational basis for the technology revolves around electrical current flowing through the muscle can be used to activate the muscle.

#### 2.1.3 Device Overview

FIGURE 1: SYSTEM SPECIFICATIONS

| Frequency | Up to 4khz |
|----------------------------|-----------------------------------------------|
| Output power | Up to a 100mA |
| Number of Electrodes | 8 electrodes with disposables contact pads |
| Simulation | Biphasic and Interferential Waveforms |
| Pulse Repetition Rate | Up to 200Hz |
| Pulse Width | Up to 290 us |
| Handpieces/Delivery System | Single use Hydrogel electrode Round or Square |

## 2.2 RATIONALE

In accordance with the definition of "Significant Risk Device" provided in 21 CFR 812.3, the devices to be used in this study has been determined to be a Non-Significant Risk device based on the following:

- a) It is not an implant
- b) It is not purported or represented to be for use in supporting or sustaining human life and do not present a potential for serious risk to the health, safety or welfare of a subject
- c) It is not for a use of substantial importance in diagnosing, curing, mitigating, or treating disease or otherwise preventing impairment of human health
- d) Use of the device does not pose a serious risk to the health, safety, or welfare of a subject.

## 2.3 POTENTIAL RISKS AND BENEFITS

## 2.3.1 Known Potential Risks

Expected adverse events of the muscle Electrical stimulation treatment procedure include:

- Transient tenderness
- Erythema
- Edema
- Discomfort

Other adverse events may include and include:

- Localized tenderness
- Skin burn
- Hyperpigmentation
- Hypopigmentation
- Blister
- Changes in skin laxity (rarely, skin contour irregularities, dimpling, and asymmetry).

Risks will be mitigated by conducting this protocol with an investigator experienced in the therapeutic area of the clinical investigation. The investigator will be trained by the sponsor on the use of the device. The device design incorporates safety mechanisms which minimize risks. Patients will also be rigorously screened prior to their enrollment and rigorously followed over the course of the study.

#### 2.3.2 Contraindications

Do not use this device on the pectoral area or patients who have a cardiac pacemaker, implanted defibrillator or other implanted metallic or electronic device. Do not use this device on patients whose pain syndromes are undiagnosed. Avoid direct irradiation of the eyes. Do not treat locally over the endocrine glands. Do not treat ischemic tissues in individuals with vascular disease.

#### 2.3.3 Known Potential Benefits

If the subject agrees to participate in this study, he/she will be contributing to the understanding of the safety and efficacy of the use of this investigational device for muscle toning. This understanding may lead to optimization of the treatment with this device.

## OBJECTIVES AND PURPOSE

## 3.1 STUDY OBJECTIVES

The objective of this clinical study is to assess the safety and efficacy of using a non-invasive electrical stimulation system for circumferential reduction and improvement of muscle strength and muscle tone of the core and extremities.

## 3.2 STUDY ENDPOINTS

## 3.2.1 Primary Endpoint

 Photographic evaluation by an independent, blinded reviewer with correct identification of pretreatment baseline images when compared to post-treatment images taken at follow up visits (30 days, 90 days). Results will be reported as a % of the correctly identified post treatment photographs chosen per Blinded Reviewer. An average of the % of the correctly identified post treatment photographs chosen by Blinded Reviewer will be calculated and used to determine efficacy.

Bar, pie charts or graphs indicating percentages of the correctly identified post treatment photographs chosen by Blinded Reviewer may also be used to analyze efficacy.

## 3.2.2 Secondary Endpoints

The secondary endpoints of this clinical trial include:

- 1. Improvement in muscle strength of the treated extremity as measured by a dynamometer at follow up visits compared to baseline measurements.
- 2. Reduction in circumference as measured by Seca Circumferential System at follow up visits compared to baseline measurement.
- 3. To assess subject satisfaction using Satisfaction Survey at each follow up visit
- 4. GAIS (Global Aesthetic Improvement Scale) by Expert Clinician.
- 5. All statistical tests that will be two-sided. The level of statistical significance for effectiveness analyses is 5% ( $\alpha$  = 0.05) for all tests of differences. Where appropriate, two-proportion z-test will be used to compare the subjects' assessment of satisfaction at post-treatment visits. Analysis of Covariance (ANCOVA) may also be used where appropriate.

## STUDY DESIGN AND ENDPOINTS

## 4.1 DESCRIPTION OF STUDY

Open-label, baseline-controlled, multi-center study evaluating an electrical muscle stimulation system for circumferential reduction and improvement in muscle strength and muscle tone of the core and extremities. The study will enroll up to 60 subjects desiring circumferential reduction and to improve muscle strength and muscle tone of their core and extremities. Each subject will receive up to 8 biweekly treatments over a 4-week period. Follow up visits planned for 30- and 90-days post treatment. Measurement outcomes will be compared to baseline.

#### 4.2 DURATION OF STUDY

This study is not expected to exceed 12 months in duration.

## SUBJECT ENROLLMENT AND WITHDRAWAL

## 5.1 Participant Improvement Criteria

The study population will consist of males and females aged 18 - 60 years of age who have chosen to participate in this clinical trial as evidenced by execution of the informed consent document.

#### 5.1.1 Informed Consent

Written informed consent will be obtained from all subjects before any study-related procedures, including any pre-treatment screening procedures, are performed. Investigators, or delegated study personnel, may discuss the availability of the study and the possibility for entry with a potential subject without first obtaining consent. Informed consent must be obtained and documented prior to initiation of any procedures that are performed solely for the purpose of determining eligibility for research.

Investigators have ethical and legal responsibilities to ensure that the protocol is clearly explained to each subject considered for enrollment in the study. Compliance with this requirement should be documented on a written Informed Consent Form approved by the reviewing IRB. Each Informed Consent Form will include the elements required by FDA regulations in 21 CFR Part 50.

The IRB-approved Informed Consent Form will be signed by the study personnel obtaining consent. The subject will be given a copy of the signed Informed Consent Form. The investigative site will keep the original on file.

## 5.1.2 Pre-treatment Recruiting/Screening

Subjects will be recruited from the study site's patient database or IRB approved advertisement and screened. Study site personnel will explain the design and purpose of the study to potential study subjects. Subjects interested in participating will visit the study site where informed consent will be obtained.

## 5.1.2.1 Screen Failures

A screen failure subject is one from whom informed consent is obtained and is documented in writing (i.e., subject signs an Informed Consent Form), but who does not receive a test spot exposure visit because of failure to meet all the eligibility criteria. Screen failure subjects will be included in the total number of subjects enrolled (i.e., all subjects consented), but not counted towards the total subjects treated.

## 5.1.3 Inclusion Criteria

Subjects must meet all the following criteria for study enrollment:

- Able to read, understand and voluntarily provide written informed consent.
- 2. Healthy male or female, ≥ 18 years to 60 years of age seeking treatment for circumferential reduction and improvement of muscle strength and muscle tone in the core and extremities.
- 3. Subject is determined to be physically fit and agrees to not making any major changes in their diet or lifestyle during the study.
- 4. Able and willing to comply with the treatment/follow-up schedule and requirements.
- 5. Women of child-bearing age are required to be using a reliable method of birth control at least 3 months prior to study enrollment and for the duration of the study and have a negative Urine Pregnancy test at baseline.

## 5.1.4 Participant Exclusion Criteria

Subjects will be excluded if they meet any of the following criteria:

- 1. Pregnant in the last 3 months, intending to become pregnant, postpartum or nursing in the last 6 months.
- 2. Any previous liposuction/lipo-sculpture or any type of surgical procedure in the treatment area in the past 12 months.
- 3. History of immunosuppression/immune deficiency disorders (including AIDS and HIV infection) or use of immunosuppressive medications, 6 months prior to and during the study.
- 4. History of hyperlipidemia, diabetes mellitus, hepatitis, blood coagulopathy or excessive bleeding.
- 5. Having a history of skin cancer or any other cancer in the areas to be treated, including presence of malignant or premalignant pigmented lesions.
- 6. Having a permanent implant in the treatment area such as metal plates or an injected chemical substance such as silicone in the treatment area.
- 7. Suffering from significant skin conditions in the treatment area or inflammatory skin conditions including but not limited to open lacerations, abrasions, herpes sores, cold sores, active infections.
- 8. Poor skin quality (severe laxity).
- 9. Abdominal wall, muscular abnormality or hernia on physical examination.
- 10. As per the investigator's discretion, any physical or mental condition which may make it unsafe for the subject to participate.
- 11. Unable or unlikely to refrain from sun exposure, artificial tanning, including the use of tanning booths, prior to 6 weeks and during the duration of the study.
- 12. Subjects unwilling or unable to adhere to all study requirements for treatment and follow-up
- 13. Investigator may exclude any subject at any time at his/her discretion

After subjects have provided informed consent and met the inclusion/exclusion criteria, the study procedures described in the following section will be performed.

## 5.2 STRATEGIES FOR RECRUITMENT AND RETENTION

Subjects will be recruited from the site's patient database and surrounding area. Site personnel should conduct/send reminder phone calls, emails, and/or text messages to remind subjects of upcoming appointments. The next appointment should be scheduled prior to the subject leaving the current appointment.

All subjects who have signed an Informed Consent Form, except for screen failures, will be considered enrolled in the study. Subjects who complete the study duration will be considered to have completed the study. Any subject who does not return for a scheduled follow-up visit will be contacted at least twice by telephone to determine the cause for the missed visit and to try to get the subject scheduled for the follow-up. A new visit will be scheduled as soon as possible. All subjects should be followed until completing the study follow-up or until study discontinuation (withdrawal) for other reasons. The reason for study discontinuation should be documented for each subject. Subjects will be deemed "Lost-to-Follow-up" if they have not returned within six weeks after the last follow-up target. For any subject lost to follow-up at least three attempts to contact the subject must be documented; the attempts must be two phone calls/emails and a registered letter.

#### 5.2.1 Subject Payment

Subjects will not be compensated for participation in this study.

## 5.3 Participant Withdrawal and Termination

All subjects have the right to withdraw at any point during the study without prejudice. The investigator can discontinue any subject, at any time, if medically necessary. Subjects must be discontinued from the investigation by the investigator at any time for any of the following reasons:

- 1. Withdrawal of informed consent.
- 2. Pregnancy (no further study-related treatments will be performed; however, the follow-up visit will be completed if the study treatments has been completed and the subject will be followed to term, called after the pregnancy, childbirth, and/or pregnancy termination and queried for abnormalities or complications).
- 3. Any AEs for which treatment continuation would constitute an unacceptably high risk for the subject.

The reason for any subject's withdrawal should be documented on the appropriate study-specific data form.

## 5.4 Premature Termination or Suspension of the Study or Study Site

The study or study site can be prematurely terminated or suspended by the sponsor. Reasons for termination of the study or a study site may include, but are not limited to, the following:

- 1. Subject enrollment is unsatisfactory.
- 2. The risks and benefits of continuing the study have been reassessed, and the risks outweigh any potential benefits.
- 3. The incidence of AEs constitutes a potential health hazard to the subjects.
- 4. New scientific data do not justify a continuation of the study.
- 5. The investigator or study site exhibit serious and/or persistent non-adherence to the protocol, the Declaration of Helsinki, EN ISO 14155, and/or applicable regulatory requirements.
- 6. The sponsor decides to terminate the study at any time for any other reason.

Furthermore, the study may be prematurely ended if the regulatory authority or the IRB has decided to terminate or suspend approval for the study, the study site, or the investigator.

If the study is prematurely terminated or suspended for any reason, the investigator must inform the subjects and assure appropriate follow-up treatment. Within the timeframes noted in applicable regulations, the sponsor will promptly inform the investigators, study sites, the IRB, and regulatory authorities of the termination or suspension of the study, as well as provide reasons for the action.

## STUDY PROCEDURES AND SCHEDULE

## 6.1 PHOTOGRAPHY

Standardized baseline and follow-up images will be taken as per specified Photography Procedure. A checklist is included in CRF to ensure "Standardized Images" are taken at specified visits. A series of standardized high-resolution digital photographs and/or video will be taken before and after treatment under controlled position and lighting conditions. Subjects will dress comfortably in loose garments and will be provided with disposable undergarments for photographs.

Prior to Taking Photographs:

- 1. Jewelry Removed
- 2. Disposable undergarments will be supplied

## While Taking Photographs

1. Photographer will position subject for photographs

#### LABORATORY EVALUATION

After Taking Photographs (before subject leaves the office)

- 1. Ensure all views have been taken
- 2. Ensure all photographs are in focus
- 3. Ensure lighting is consistent

## 6.2 STUDY SCHEDULE

## 6.2.1 Study Specific Procedures

The following procedures will be done as part of this study:

- 1. Demographics (Visit 1)
- 2. Medical/surgical history
- 3. Concomitant medications
- 4. Assessment of eligibility (inclusion/exclusion criteria)
- 5. Urine pregnancy test for women of child-bearing potential (Visit 1 only)
- 6. Adverse event reporting
- 7. Photography (Pre-treatment, post-treatment and at follow up visits)
- 8. Weight and circumferential measurements (Visit 1 and follow up visits only)
- 9. Dynamometer measurements (Visit 1 and follow up visits only)
- 10. Subject Satisfaction Survey (at follow up visits only)

## 6.3 LABORATORY EVALUATION

Women of child-bearing potential will be asked to provide a urine sample for a urine pregnancy test to be performed according to local site standards. Urine pregnancy required within 24 hours of study intervention. A negative result must be available prior to administration of the treatment.

A staff member will explain how the pregnancy test will be performed at the screening visit depending on which type of pregnancy test is available at the study center. Instructions will include:

- 1. Hold the pregnancy test stick directly under your urine for 5-10 seconds.
- 2. Alternatively, you may be asked to urinate into a specimen cup and dip the pregnancy test stick into the urine for 5-10 seconds.
- 3. Results are typically available within 2-5 minutes, but some tests take as long as 10 minutes.
- 4. A positive result indicating pregnancy will usually be a colored line or plus symbol in the result window. A negative result indicating no pregnancy will usually be absence of a colored line or a negative symbol.

## 6.4 SCREENING AND BASELINE (VISIT 1)

The Principal Investigator or his/her designee will assess the subject eligibility for participation in the clinical study using the inclusion/exclusion criteria (Sections 5.1; 5.2). Subjects meeting the study criteria for enrollment will be asked to sign an informed consent document. The Principal Investigator or his/her

designee will obtain informed consent from the subject. All subjects must clearly indicate his/her understanding of the requirements and possible risks involved with study participation. Once subjects sign the informed consent document, they will be assigned a unique identifying number that will be composed of a two-digit site number and a three-digit subject number in sequence. This unique identifier will be used throughout the entire study and will be entered in the subject's case report form (CRF).

During the screening visit, the Principal Investigator or his/her designee will review the subjects medical/surgical history, demographic information, concomitant medication and examine the treatment area. Weight and circumferential measurements of the core and extremities.

Women of child-bearing potential will be asked the date of their last menstrual cycle and required to provide a urine sample for a urine pregnancy test. A negative result is required within 24 hours of treatment for participation in study. The investigator will inquire about contraceptive use to confirm they meet the inclusion criteria.

- 1. Obtain informed consent of potential participant verified by signature on study informed consent form.
- 2. Verify all preliminary/screening inclusion/exclusion criteria are met.
- 3. Document medical history.
- 4. Obtain pregnancy screen (if applicable).
- 5. Document concurrent medications.
- 6. Obtain demographics.

## 6.5 STUDY TREATMENT

## 6.5.1 Subject Preparation for Study Treatment

The investigator, sub-investigator, or delegated clinician will first identify the skin areas to which treatment/exposure is to be performed. Treatment records will be maintained in accordance with this protocol. Skin in the treatment area should be clean. Subject will be instructed to avoid lotion or oil on the treatment area 24 hours prior to treatment.

## 6.5.2 Study Treatment (Visits 1-8)

All study treatments will be performed by the investigator, sub-investigator, or delegated clinician (i.e., study exposure clinician as designated by the principal investigator.) The investigator will confirm that the subject continues to meet the inclusion criteria and none of the exclusion criteria prior to each study treatment. Concomitant medications will be reviewed. Specific treatment parameters will be determined by the Investigator and recorded on the case report forms.

Each subject will receive up to **8** study treatments over a **4**-week period. Subjects return for a 30 day and 90-day post final treatment follow up visit.

- Cleanse skin.
- Obtain digital images.
- Perform study treatment.
- Obtain Numeric Pain Rating Scale score.
- Assess for expected treatment effects (ETEs) and adverse events (AEs).

Subjects will be asked to return for follow up visits post-final treatment at 30 days and 90 days. At 1<sup>st</sup> and all follow up visits weight, dynamometer measurements, circumferential measurements, subject satisfaction survey, adverse events and photography will be completed and assessed.

Subject discomfort during study treatment will be documented using a 0 (None) to 10 (Severe) numeric pain rating scale. If the treatment becomes too uncomfortable for a subject, it will be discontinued, or the settings may be lowered to a more comfortable level. Subjects may also request that treatment be discontinued at any time, for any reason.

## 6.5.3 Acute Responses

For all exposures, acute responses (e.g., erythema or edema) will be observed by the study exposure clinician and recorded after exposure. If any Serious Adverse Events (SAE) are noted, an SAE Form should be completed.

## 6.5.4 Post- Care Instructions

Following treatment subject may assume normal activities. Hot baths, sauna and vigorous exercise should be avoided. The subject should be reminded to not make any major changes in their diet or lifestyle during the study.

## 6.5.5 Schedule of Activities

**TABLE 1: SCHEDULE OF ACTIVITIES** 

| TABLE 1: 3CHEDULE O | ACTIVITIES | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | FU 30 | FU 90 |
| | Screening | Tx 1 | Tx 2 | Tx 3 | Tx 4 | Tx 5 | Tx 6 | Tx 7 | Tx 8 | day | days |
| Informed | | | | | | | | | | | |
| Consent | x | | | | | | | | | | |
| Pregnancy | | | | | | | | | | | |
| Verification | x | | | | | | | | | | |
| Concomitant | | | | | | | | | | | |
| Medications | х | x | х | х | x | x | х | х | х | х | х |
| Medical History | х | | | | | | | | | | |
| Demographics | х | | | | | | | | | | |
| Weight | х | | | | | | | | | х | х |
| Dynamometer | | | | | | | | | | | |
| Measurements | х | | | | | | | | | х | х |
| Circumferential | | | | | | | | | | | |
| Measurements | x | | | | | | | | | х | х |
| Photography | | | | | | | | | | | |
| (pre- and - post | | | | | | | | | | | |
| treatment) | | x | | | | | | | | х | х |
| Subject | | | | | | | | | | | |
| Satisfaction | | | | | | | | | | х | х |

| Pain Scale Rating | | x | x | x | x | х | х | х | | |
|-------------------|---|---|---|---|---|---|---|---|---|---|
| Adverse Events | x | х | х | х | х | х | х | х | х | х |

## 6.5.6 Safety Assessments

Assess for adverse events immediately post-treatments and at the follow-up visits.

#### 6.5.7 Unscheduled Visit

Any unscheduled visit or examine should be documented in the subject's medical record and adverse event form (if applicable) stating the reason for the visit and any actions taken. The Sponsor should be notified of the unscheduled visit.

#### 6.6 STUDY TREATMENT

This study involves up to 8 treatments to be conducted after obtaining informed consent, screening for inclusion/exclusion, complying with standardized photography requirements, and completing pregnancy tests, if applicable.

#### 6.6.1 Subject Preparation for Study Treatment

The investigator, sub-investigator, or delegated clinician will first identify the skin areas to which treatment/exposure is to be performed. Treatment records will be maintained in accordance with this protocol. Skin in treatment area should be clean. No lotion or oil should be present on the area to be treated.

## 6.6.2 Study Treatment

All study treatments will be performed by the investigator, sub-investigator, or delegated clinician (i.e., study exposure clinician as designated by the principal investigator.)

Specific treatment parameters will be determined by the Investigator and recorded on the case report forms. Subject discomfort during study treatment will be documented using a 0 (None) to 10 (Severe) pain rating scale. If the treatment becomes too uncomfortable for a subject, it will be discontinued, or the settings may be lowered to a more comfortable level. Subjects may also request that treatment be discontinued at any time for any reason.

#### 6.6.3 Acute Responses

For all exposures, acute responses (e.g., erythema or edema) will be observed by the study exposure clinician and recorded after exposure. If any Serious Adverse Events (SAE) are noted, an SAE Form should be completed.

#### 6.6.4 Post- Care Instructions

Following treatment subject may assume normal activities. Hot baths, sauna and vigorous exercise should be avoided. The subject should be reminded to not make any major changes in their diet or lifestyle during the study.

## 6.7 CONCOMITANT MEDICATIONS

All concomitant prescription medications taken during study participation will be recorded on the appropriate study-specific data form. For this protocol, a prescription medication is defined as a medication that can be prescribed only by a properly authorized/licensed clinician. Medications to be

reported on the data form and entered on the CRF are concomitant prescription medications, over-the-counter medications and non-prescription medications.

## ASSESSMENT OF SAFETY

## 7.1 Specifications of Safety Parameters

## 7.1.1 Definition of an Expected Treatment Effect (ETE) and an Adverse Event (AE)

An expected treatment effect is defined as any typical treatment side-effect of the study devices of mild to moderate severity and lasting up to a typical maximum duration. An adverse event is defined as any new medical problem, or exacerbation of an existing problem, experienced by a subject while enrolled in the study, whether it is considered device-related by the investigator. All ETEs and AEs will be collected during the conduct of this trial.

## 7.1.2 Definition of Serious Adverse Event (SAE)

Each adverse event should be assessed for its seriousness. The definition below should be used for this assessment. Please note that the term serious adverse event is not synonymous with a "severe" adverse event, which may be used to describe the intensity of an event experienced by the subject.

An adverse event should be classified as serious if it meets any of the following criteria:

- a. Death
  - Death was an outcome of the adverse event.
- b. Life-threatening
  - The subject was at substantial risk of dying at the time of the adverse event or use or continued use of the device.
- c. Hospitalization (initial or prolonged)
  - Admission to the hospital or prolongation of hospitalization was a result of the adverse event.
- d. Disability or Permanent Damage
  - The adverse event resulted in a substantial disruption of a person's ability to conduct normal life functions, i.e., the adverse event resulted in a significant, persistent or permanent change, impairment, damage or disruption in the patient's body function/structure, physical activities and/or quality of life.
- e. Congenital Anomaly/Birth Defect
  - Exposure to a medical product prior to conception or during pregnancy may have resulted in an adverse outcome in the child.
- f. Required Intervention to Prevent Permanent Impairment or Damage (Devices)
  - Medical or surgical intervention was necessary to preclude permanent impairment of a body function, or prevent permanent damage to a body structure, either situation suspected to be due to the use of a medical product.
- g. Other Serious (Important Medical Events)
  - The event does not fit the other outcomes, but the event may jeopardize the subject and may require medical or surgical intervention (treatment) to prevent one of the other outcomes.

Non-serious adverse events are all events that do not meet the criteria for a "serious" adverse event.

## 7.1.3 Definition of Unanticipated Adverse Device Effects (Events)

An unanticipated adverse device effect is defined as "any serious adverse effect on health or safety, or any life-threatening problem, or death caused by, or associated with, a device; if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan,

or application (including supplementary application), or any other unanticipated serious problem associated with a device that relates to the rights, safety, or welfare of subjects."

## 7.2 CLASSIFICATION OF AN EVENT

## 7.2.1 Severity of Event

Each adverse event should be assessed for its severity, or the intensity of an event experienced by the subject, using the following classifications:

1 = Mild Discomfort noticed, but no disruption to daily activity

2 = Moderate Discomfort sufficient to reduce or affect normal daily activity

3 = Severe Inability to work or perform normal daily activity

## 7.2.2 Relationship to the Investigational Device

The investigator should assess the relationship of the adverse event to the investigational device. The relationship should be assessed using the categories presented in **Table 2**.

TABLE 2: RELATIONSHIP BETWEEN ADVERSE EVENTS AND INVESTIGATIONAL DEVICE

| Definite | Definite relationship exists between the device/procedure and an adverse event |
|---|---|
| Probably Related | A reasonable causal relationship between the device/procedure and an adverse event is more likely than not. |
| Possibly Related | A reasonable relationship exists between the device/procedure and an adverse event, but the causal relationship is unclear or lacking. |
| Not Likely Related | A temporal relationship exists between the device/procedure and an adverse event, but there is no reasonable causal relationship. For example, the adverse event occurs in a time frame, which makes a causal relationship to device treatment improbable. |
| Unrelated | No relationship between treatment with the device/procedure and the adverse event exists. |

#### 7.2.3 Expectedness

Reported events will be categorized as Expected Treatment Effects if the event meets the definition of any typical treatment side-effect of study devices of mild to moderate severity and lasting up to a typical maximum duration.

## 7.3 TIME PERIOD AND FREQUENCY FOR EVENT FOLLOW UP AND ASSESSMENT

The occurrence of an AE or SAE may come to the attention of study personnel during a study visit or upon review by a study monitor. All ETEs and AEs will be captured on the appropriate data form. Information to be collected includes event description, date of onset, clinician's assessment of seriousness and severity, relationship to study device/treatment (assessed only by those with the training and authority to decide), actions taken, and date of event resolution. All AEs occurring while on study must be documented appropriately regardless of relationship. All ETEs/AEs assessed as "not yet resolved" must continue to be followed via telephone contact, email or clinic visit every 7 days or sooner as per the physician's direction until event resolution or stabilization or tissue resection.

A pre-existing condition should not be reported as an adverse event unless there has been a substantial increase in severity or frequency of the problem that has not been attributed to natural history.

Changes in the severity of an event will be documented to allow for a determination if the event should be re-categorized from an ETE to AE.

The PI will record all reportable events with start dates occurring any time after informed consent is obtained until 7 (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation or until tissue is resected. At each study visit, the investigator will inquire about the occurrence of ETEs/AEs/SAEs since the last visit. Events will be followed for outcome information until resolution or stabilization or tissue is resected.

## 7.4 Reporting Procedures

#### 7.4.1 Adverse Event Reporting

Any new medical problem, or an exacerbation of an existing condition, reported from the time the informed consent form is signed must be followed until the last study visit after the last study treatment/exposure or until event resolution.

AEs will not be followed up after the final study visit as tissue will be resected at the abdominoplasty visit. AEs related to the abdominoplasty are outside the scope of this study and will not be reported.

#### 7.4.2 Serious Adverse Event Reporting

Serious adverse events must be reported to the Sponsor as soon as possible, preferably within 24 hours but in no event later than 72 hours. Any AE considered serious by the PI or Sub-investigator or which meets the definition of an SAE included in **Section 7.1.2, Definition of Serious Adverse Event** must be documented on an SAE data form.

The Sponsor will conduct an investigation. If the Sponsor determines that the investigation presents an unreasonable risk to subjects, all investigations or parts of the investigation presenting that risk will be terminated as soon as possible. The investigator must report serious adverse events to the reviewing IRB according to the IRB regulations at the study site.

## 7.4.3 Unanticipated Adverse Device Effect Reporting

If an unanticipated adverse device effect occurs, the study investigator shall complete the appropriate study-specific data form and submit to the study sponsor and to the reviewing IRB as soon as possible, but in no event later than 10 working days after the investigator first learns of the effect. The study sponsor contact information is provided in **Section 1**, **Key Roles**. The study sponsor is responsible for conducting an evaluation of an unanticipated adverse device effect and shall report the results of such evaluation to FDA and to all reviewing IRBs and participating investigators within 10 working days after the sponsor first receives notice of the effect. Thereafter the sponsor shall submit such additional reports concerning the effect as FDA requests.

#### 7.4.4 Reporting of Pregnancy

Each pregnancy that starts during the subject's study participation must be reported by the investigator to the Sponsor within 24 hours of learning of its occurrence. Pregnancies and pregnancy follow-up should be reported on an Adverse Event form. Pregnancy follow-up should describe the outcome of the pregnancy, including any voluntary or spontaneous discontinuation; details of the birth; the presence or absence of any congenital abnormalities, birth defects, maternal or newborn complications, and their relation to the device or treatment/exposure. Each pregnancy must be reported as a non-serious AE if the subject has received at least one study treatment/exposure. The following criteria should be followed:

- a. If a subject becomes pregnant after the Baseline visit and all study treatments/test spot exposure have been completed, the subject should continue to be followed for the duration of the pregnancy.
- b. If a subject becomes pregnant after the Baseline visit but before any study treatments/test spot exposures, the subject should be exited from the study.
- c. If a subject becomes pregnant after the Baseline visit but before all study treatments/test spot exposures have been completed, additional study treatments/test spot exposures should be discontinued, and the subject should continue to be followed for the duration of the pregnancy.

#### 7.4.5 Reporting of Deaths

The investigator must notify the Sponsor as soon as possible, preferably within 24 hours but in no event later than 48 hours, of learning of a subject's death, regardless of whether the death is related or unrelated to the investigational device. The investigator should attempt to determine, as conclusively as possible, whether the death is related to the device. The cause of death and the investigator's discussion regarding whether the death was device-related should be described in a written report. The investigator mush report death to the reviewing IRB according to the IRB regulations at the study site.

## 8. CLINICAL MONITORING

Clinical site monitoring is conducted to ensure that the rights and well-being of human subjects are protected, that the reported trial data are accurate, complete, and verifiable, and that the conduct of the trial is in compliance with the currently approved protocol/amendment(s), with GCP, and with applicable regulatory requirement(s).

- 1. Monitoring for this study will be performed by the Sponsor or Sponsor contract monitor.
- 2. Clinical study site and data monitoring will be conducted via both centralized and on-site monitoring.
  - a. Centralized data monitoring will focus primarily on:
    - i. Ongoing, real-time review of clinical data supporting safety, and primary and secondary study-defined endpoints, specifically:
      - 1. Tracking the occurrence of adverse events and expected treatment effects.
    - ii. Ongoing, real-time review of clinical data as entered on Case Report Forms (CRF):
      - 1. Initial study consent was obtained for all enrolled subjects;
      - 2. Eligibility for study participation of all enrolled subjects;
      - 3. Verification of protocol compliance and data completeness.
    - iii. Ongoing, real-time evaluation of data trends to identify outliers, unexpected trends, or holes in data collection;
    - iv. Ongoing, real-time evaluation of study photographs.
  - b. Centralized monitoring requires timely data entry and timely uploading of completed CRFs to the study HIPAA compliant cloud-based system, e.g., no later than 7 working days after a study visit has occurred.
  - c. On- site monitoring visits will include:
    - i. Review of primary/secondary endpoint data source documents;
    - ii. Confirmation that subject randomization is being completed appropriately (if applicable);
    - iii. Confirmation that study blinding is maintained (if applicable);

- iv. Confirmation of appropriate execution of the PGAIS, SGAIS, PSQ, or other study-specific scales;
- v. Note any other study-specific study design items requiring on-site confirmation.
- d. General on-site monitoring tasks will include:
  - i. Review of study conduct and progress at each investigative site, e.g., protocol compliance, subject recruitment, etc.;
  - ii. Confirmation that written informed consent was obtained and documented at the time of screening, using an appropriate version of an IRB-approved ICF, and subject eligibility is confirmed.
  - Confirmation that all expected treatment effects, adverse events and/or protocol deviations noted in site records are appropriately documented on study specific CRFs.
  - iv. Identification and resolution of any device performance issues;
  - v. Review of the investigator's study records, study management documents and subject informed consent documents.
  - vi. Confirmation that all investigative site personnel with study-related responsibilities are adequately trained and that the applicable training records are maintained in the Site Regulatory Binder.
  - vii. Confirmation that study-related responsibilities of site personnel are appropriately documented on the Delegation of Responsibility Log and the log is maintained in the Site Regulatory Binder.
  - viii. Reconciliation of the Device Disposition Log against device inventory and confirmation that study devices are kept in a secure location.
  - ix. Confirmation that required regulatory documents are present in the Site Regulatory Binder and are current and correct.
  - x. Ensure that all findings, conclusions and any actions taken to correct deficiencies noted during an on-site monitoring visit are documented in a site monitoring report.
- e. On-site monitoring frequency
  - i. An on-site monitoring visit will be completed at each study site at least one time during this clinical trial.
  - ii. The frequency of site monitoring visits may be adjusted based on a number of factors, including but not limited to:
    - 1. Duration of the study;
    - 2. Number of subjects enrolled;
    - 3. Number of investigators/sites;
    - 4. Complexity of the study;
    - 5. The level of the study site's experience in conducting and overseeing clinical trials;
    - 6. The quality of the data documented on study-specific data forms and entered into the study database;
    - 7. Number of outstanding issues from previous visits.

## 9. STATISTICAL ANALYSIS

## 9.1 STATISTICAL AND ANALYTICAL PLANS

The primary analysis of efficacy will be based on the evaluable treated subjects, hence, only those subjects who received complete study treatments and follow up visits will be included in the analysis.

#### 9.2 Analysis Datasets

The following analysis sets will be defined for the statistical analysis of this investigation:

#### Safety Evaluation Set (SES)

Subset of all subjects who received the investigational treatment.

#### Full Analysis Set (FAS)

Subset of subjects in SES that received complete treatments have primary effectiveness data available.

## Per Protocol Set (PPS)

Subset of all subjects who received complete treatments and have completed the study without major protocol deviations.

## 9.3 Description of Statistic Methods

Endpoints will be summarized using descriptive statistics including mean score, standard deviation, standard error and range. Frequency and percentage of subjects within each category will be presented for categorical data. If applicable, Wilcox t-test may be used to determine if two sets of data are significantly different from one another. If p-value is below the level of statistical significance for effectiveness analyses ( $\alpha$  = 0.05) for all tests of differences, then the null hypothesis is rejected in favor of the alternative hypothesis. Rejection of null hypotheses will establish that:

- The two-sided 95% confidence interval for the difference between the means excludes zero.
- The two means are statistically significantly different at the 5% level (P < 0.05) two-sided</li>

Upon rejection of null hypotheses, further statistical test tools such as, Confidence Interval, and/or One-way ANOVA and/or descriptive statistical tools may be used to determine the performance of the treatment.

#### 9.4 SAFETY ANALYSES

The safety analysis will be done by analyzing spontaneous reports of adverse events (AE), as well as analysis of immediate response reports by the principal investigator from his/her observation/examination of the treated area. Appropriate Medical Dictionary for Regulatory Activities (MedDRA) code will be used to describe all spontaneously reported events or other study related adverse events.

Summaries of spontaneously reported or other study related adverse events will be presented as:

- Number (%) of subjects with any AE
- Number (%) of subjects with any serious adverse events (SAE)
- Number (%) of subjects permanently withdrawn from treatment due to AE

Summaries of analysis of immediate response reports by the principal investigator examination will be displayed on a bar or pie chart and/or a table as;

- a. The overall frequency of subjects with each event (pain during treatment, hemorrhage, burn, erythema, edema, purpura, etc.).
- b. Frequency of subjects with specific severity/intensity for each event using a 5-pointscale: 1=none; 2=trace; 3=moderate; 4=marked; 5=severe.

c. The overall proportion of subjects observed with marked or severe intensity of any event will be calculated and compared to those with none, trace or moderate severity/intensity.

## 9.6 Baseline Descriptive Statistics

Subjects' baseline demographics will be compared using descriptive statistics such as mean score, standard deviation, standard error and range. Data will be displayed in tables or graphical presentation.

#### 9.7 ANALYSIS OF PRIMARY ENDPOINTS

The following will be considered for the analysis of primary endpoints:

The results of each Blinded Reviewer's evaluation of photographs taken at 1 month and 3 months compared to baseline will be analyzed, and the results will be reported as a % of the correctly identified post treatment photographs chosen per Blinded Reviewer. An average of the % of the correctly identified post treatment photographs chosen by Blinded Reviewer will be calculated and used to determine

Bar, pie charts or graphs indicating percentages of the correctly identified post treatment photographs chosen by Blinded Reviewer may also be used to analyses efficacy.

The % of the correctly identified post treatment photographs chosen by Blinded Reviewer of all subjects who received all treatments with the investigational device and for whom all valid post-baseline assessment was obtained will be analyzed for these primary endpoints. Multiple imputation method or modelling of available data may be used for missing data as appropriate.

#### 9.8 Analysis of Secondary Endpoints

For the analysis of changes in muscle tone and muscle strength, circumference of the extremities and subjects' assessment of satisfaction with the treatment secondary endpoints, the following analysis will be considered:

Summary tables of changes in measurements of muscle tone and strength, circumference and subjects' assessment of satisfaction at 1 and 3 months post last treatment as compared to baseline will be displayed as mean difference, standard deviation and standard error.

Bar charts, pie chart, graphs or any other descriptive statistical displays indicating scores, percentages and/or proportions of changes in circumference and subjects' assessment of satisfaction at 1 month and 3-month post-treatment as compared to baseline will be used where applicable to analyze efficacy.

All statistical tests that will be two-sided. The level of statistical significance for effectiveness analyses is 5% ( $\alpha$  = 0.05) for all tests of differences. Where appropriate, two-proportion z-test will be used to compare the differences between changes in abdominal circumference and subjects' assessment of satisfaction at 1 month and 3 months post last treatment as compared to baseline.

Analysis of Covariance (ANCOVA) may also be used where appropriate. Change in abdominal circumference and subjects' assessment of satisfaction assessments at twelve weeks post-treatment as compared to baseline of all subjects who received all treatments with the investigational device and for whom have all valid post-baseline assessment was obtained will be analyzed for these secondary

endpoints. Multiple imputation method or modelling of available data may be used for missing data as appropriate.

## 10. SOURCE DOCUMENTS AND ACCESS TO SOURCE DOCUMENTS

Source documents are defined as the results of original observations and activities of a clinical investigation. Source documents will include, but are not limited to, study-specific data forms, progress notes, electronic data, computer printouts, screening logs, and recorded data from automated instruments. All source documents pertaining to this study will be maintained by the investigators and made available for inspection by authorized persons.

Following written SOPs, the clinical study monitors will verify that the clinical trial is conducted, and data are generated, documented (recorded), and reported in compliance with the protocol, GCP, and the applicable regulatory requirements.

The investigational site will provide direct access to all trial related sites, source data/documents, and reports for the purpose of monitoring and auditing by the sponsor, and inspection by local and regulatory authorities.

# 11. ETHICS/PROTECTION OF HUMAN SUBJECTS

## 11.1 ETHICAL STANDARD

This clinical study will be conducted in accordance with the Protection of Human Subjects Regulations, including Subpart B Informed Consent of Human Subjects (21 CFR Part 50); the Institutional Review Board Regulations (21 CFR Part 56); the Financial Disclosure by Clinical Investigators Regulations (21 CFR Part 54); and the Investigational Device Exemptions Regulations (21 CFR Part 812), and the ICH E6.

## 11.2 Institutional Review Board

Prior to initiation of any study procedures, the protocol, informed consent, and recruitment materials, and all participant materials will be submitted to a duly constituted IRB for view and approval. In addition, any amendments to the protocol or Informed Consent Form will be reviewed and approved by the IRB. The Sponsor must receive a letter documenting IRB approval at the clinical site prior to the initiation of the study.

The investigator is responsible for providing the appropriate reports to its reviewing IRB during the clinical study. These reports will include:

- 1. Informing the IRB of the study progress periodically as required, but at least annually;
- 2. Reporting any unanticipated adverse device effects within 10 working days of first learning of the event;
- 3. Reporting any deviations from the clinical protocol to protect the life or well-being of a subject in the case of an emergency within five working days after the emergency occurred;
- 4. Reporting the use of the device without obtaining informed consent from a subject within five working days of the event; and
- 5. Providing any other reports requested by the IRB.

The IRB must be notified of study completion within 30 days of the final visit of the last subject and should be provided with a summary of the results of the study by the investigator.

#### 11.3 INFORMED CONSENT PROCESS

11.3.1 Consent/Assent and Other Informational Documents Provided to Participants Consent forms describing in detail the study device, study procedures, and risks are given to the participant and written documentation of informed consent is required prior to starting intervention/administering study product.

#### 11.3.2 Consent Procedures and Documentation

Informed consent will be obtained from all subjects prior to study participation. Informed consent is a process that is initiated prior to the individual's agreeing to participate in the study and continues throughout the individual's study participation. Extensive discussion of risks and possible benefits of participation will be provided to each participant. Consent forms will be IRB-approved, and the participant will be asked to read and review the document. The investigator, or investigator-delegated study personnel, will explain the research study to the participant and answer any questions that may arise. All participants will receive a verbal explanation in terms suited to their comprehension of the purposes, procedures, and potential risks of the study and of their rights as research participants. Participants will have the opportunity to carefully review the written consent form and ask questions prior to signing. The participants should have the opportunity to discuss the study with their surrogates or think about it prior to agreeing to participate. The participant will sign the informed consent document prior to any procedures being done specifically for the study. The participants may withdraw consent at any time throughout the course of the trial. A copy of the informed consent document will be given to the participants for their records. The rights and welfare of the participants will be protected by emphasizing to them that the quality of their medical care will not be adversely affected if they decline to participate in this study.

#### 11.4 Participant and Data Confidentiality

All information generated in this study must be considered highly confidential and must not be disclosed to any persons not directly concerned with the study without prior written permission from the Sponsor. Authorized regulatory officials and Sponsor personnel (or its representatives) will be allowed full access to inspect the records. All investigational devices and/or other materials collected will be used solely in accordance with this protocol, unless otherwise agreed to in writing by the Sponsor. Subjects should be identified only by initials and unique subject numbers on study-specific data forms. If necessary, their full names may be made known to a regulatory agency or other authorized officials.

## 12. DATA HANDLING AND RECORD KEEPING

## 12.1 Data Collection and Management Responsibilities

Data collection is the responsibility of the clinical trial staff at the site under the supervision of the site PI. The investigator is responsible for ensuring the accuracy, completeness, legibility, and timeliness of the data reported.

During each subject's visit to the clinic, study data will be documented by study personnel on study-specific data forms (CRFs). In addition, study personnel will record progress notes to document all significant observations, and any contact with a subject by telephone or other means that provides significant clinical information will also be documented in the progress notes as described above. For transmission to the Sponsor, information from the study progress notes and other source documents will be promptly transcribed to study-specific data forms (CRFs). In this clinical trial, study-

specific data forms (CRFs) may also serve as source documents. Transcription of study data onto study-specific data forms should be completed and uploaded within 7 days of the study visit.

Copies of the CRF serving as source documents must be maintained for each participant enrolled in the study. Data reported in the CRF derived from source documents should be consistent with the source documents or the discrepancies should be explained and captured in a progress note and maintained in the participant's official study record.

Any changes to information in the study progress notes, other source documents, and data forms will be initialed and dated in ink on the day the change is made by a site study staff member authorized to make the change. Changes will be made by striking a single line through erroneous data, and clearly entering the correct data. If the reason for the change is not apparent, a brief explanation for the change will be written in the source documentation by the clinician.

## 12.2 INVESTIGATOR RECORDS AND REPORTS

## 12.2.1 Investigator Records

Prior to participation in the investigation, the investigator must provide the following documentation to the Sponsor:

- Investigator Agreement, signed by the investigator, which lists any physicians who will be involved in conducting the investigation under the direction of the primary investigator;
- A copy of the principal investigator's, sub-investigator's, other delegated study clinicians' curriculum vitae;
- A letter signed by the chairperson of the IRB overseeing the conduct of this study indicating that the IRB has reviewed and approved this investigational plan; and
- A copy of the IRB-approved Informed Consent Form.
   During the study, investigators are required to maintain on file the following accurate, complete, and current records relating to this study as described in 21 CFR §812.140. A summary of these records is listed below:
- All correspondence and required reports, which pertain to the study.
- Records of receipt, use, or disposition of study devices, including the type and quantity of devices; the dates of receipt; the serial numbers; the names of all persons who received, used or disposed of each device; and why and how many units of the device have been returned to the Sponsor, repaired, or otherwise disposed.
- o Records of each subject's case history and exposure to the device.
- Signed and dated consent forms.
- Relevant observations, including records concerning adverse events, condition of each subject upon entering and results of diagnostic tests.
- Study-specific data forms and corrections to the forms.
- o Protocol and amendments.
- Subject recruiting materials.
- Investigator curriculum vitae.

## 12.2.2 Investigator Reports

Investigators are required to prepare and submit to the Sponsor the following complete, accurate, and timely reports on this investigation when are required. These reports, which are listed below, are required by 21 CFR §812.150; additional reports may be requested by the Sponsor:

• The investigator will notify the Sponsor of a subject death occurring during the investigation, as soon as possible, preferably within 24 hours of learning of the subject's death, but in no event

later than 48 hours. The investigator will notify the reviewing IRB of a subject death as specified by the IRB.

- The investigator will notify the Sponsor of any unanticipated adverse device effects within 48 hours after learning of the effect. The investigator will notify its reviewing IRB of any unanticipated adverse device effects, as soon as possible, but no later than 10 working days after learning of the effect.
- The investigator will notify the Sponsor of the withdrawal of IRB approval, as soon as possible, but no later than five working days after learning of the withdrawal.
- The investigator will provide current progress reports to the Sponsor and reviewing IRB at regular intervals and at least on an annual basis.
- The investigator will notify the Sponsor and reviewing IRB of any deviation from the investigational plan to protect the life and physical well-being of a subject in an emergency, as soon as possible, but no later than five working days after the emergency occurred.
- The investigator will notify the Sponsor and reviewing IRB that an informed consent was not obtained from a subject, as soon as possible, but no later than five working days after such an occurrence.
- The investigator will provide a final summary report to the Sponsor and reviewing IRB within three months after termination or completion of the study.
- The investigator will provide any other information upon the request of an IRB, FDA, or the Sponsor.

## 12.3 STUDY RETENTION RECORDS

The investigator is responsible for retaining the necessary records, including a copy of the protocol, device labeling, study-specific data forms, medical records, original reports of test results, all study-related correspondence, a record of written informed consent, and any other documents pertaining to the conduct of this study.

FDA regulations require all investigators participating in investigational device studies to maintain detailed clinical records during the investigation and for a period of at least two years after the latter of the following two dates:

- 1. The date on which the investigation is terminated or complete; or
- 2. The date the records are no longer required for purposes of supporting a premarket approval application.

The investigator must not dispose of any records relevant to this study without either:

- 1. Obtaining written permission from the Sponsor; or
- 2. Providing an opportunity for the Sponsor to collect such records.

The investigator shall take responsibility for maintaining adequate and accurate electronic or hard copy source documents of all observations and data generated during this study. Such documentation is subject to inspection by the Sponsor and the FDA.

## 12.4 PROTOCOL DEVIATIONS

This study should be conducted as described in this protocol, except for an emergency in which the protection, safety, and well-being of a subject requires a protocol deviation, based on the judgment of the investigator (or a responsible, appropriately trained professional designated by the investigator). If the deviation from the protocol is necessary to protect the physical well-being of a subject in an

emergency, such protocol deviations must be reported to the Sponsor and the reviewing IRB as soon as possible, but no later than five working days after the emergency occurred.

In the event of a significant deviation from the protocol due to an accident or mistake, the investigator or designee must contact the Sponsor at the earliest possible time by telephone to discuss the deviation and its impact on the study and subject continuation in the study. These discussions will be documented by the investigator and the Sponsor and reviewed by the monitor.

#### 12.5 Publication and Data Sharing Policy

The data produced by this Lutronic-sponsored study is the sole property of Lutronic. Thereby, abstracts, publications and presentations of this data must be pre-approved by Lutronic in writing (e-mail approval is acceptable). The Sponsor must also be provided with the opportunity to review all investigator-prepared abstracts, publications or presentations. A period of thirty (30) days for presentational materials and abstracts and forty-five (45) days for manuscripts will be required for review and comment by Sponsor's Clinical Research Department. These requirements acknowledge Sponsor's responsibility to evaluate such publications for their accuracy, to ascertain whether Confidential Information is being inappropriately released, to provide the Principal Investigator with information which may not yet have been available to him/her, and to provide input from co-authors regarding content and conclusions of the publication or presentation. If requested in writing by the Sponsor, the Institution will withhold publication to protect the potential patentability of any invention described therein and/or made available to fulfill regulatory requirements. Notwithstanding the foregoing, Institution agrees that if the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results from the investigators at the other study centers as a multi-center publication.

## 13. STUDY ADMINISTRATION

#### 13.1 Study Investigators

All investigators will be experienced with aesthetic treatments using a variety of accepted clinical modalities.

#### 13.2 AMENDMENT POLICY

The investigator will not make any changes to this protocol without prior written consent from the Sponsor and subsequent approval by the IRB, except if the deviation from the protocol is necessary to protect the life and physical well-being of a subject in an emergency. Such protocol deviations must be reported to the Sponsor and the reviewing IRB as soon as possible, but no later than five working days after the emergency occurred.

Any permanent change to the protocol, whether it is an overall change or a change for specific study center(s), must be handled as a protocol amendment. Any amendment to the protocol that appears indicated as the study progresses will be fully discussed by the investigator(s) and the Sponsor. If agreement is reached regarding the need for an amendment, the Sponsor will write it. The written amendment must be submitted to the chairman of the IRB identified with this responsibility. Except for "administrative amendments", investigators must await IRB approval of protocol amendments before implementing the change(s). Administrative amendments are defined to have no effect on the validity of the data or information resulting from the completion of the approved protocol, or the relationship of likely patient risk to benefit relied upon to approve the protocol; the scientific soundness of the investigational plan or protocol; and the right, safety or welfare of the human subjects involved in the investigation.

When, in judgment of the chairman of the IRB, the investigators and/or the Sponsor, the amendment to the protocol substantially alters the study design and/or increases the potential risk to the subject, the currently approved written Informed Consent Form will require similar modification. In such cases, repeat informed consent will be obtained from subjects enrolled in the study before continued participation.

## 14. CONFLICT OF INTEREST POLICY

The independence of this study from any actual or perceived influence is critical. Therefore, any actual conflict of interest of persons who have a role in the design, conduct, analysis, publication, or any aspect of this trial will be disclosed and managed. Furthermore, persons who have a perceived conflict of interest will be required to have such conflicts managed in a way that is appropriate to their participation in the trial.

## References

- Bélanger A: Therapeutic Electrophysical Agents: Evidence Behind Practice, Williams and Wilkins, A Walters Kluwer Business, 2010.
- Cohn JC and Mullin C: Neuromuscular Applications for Electrical Stimulation, from Physical Agents for the Physical Therapist Assistant, FA Davis Company, 1996.
- Gillespie CA: Foundations for Electrical Stimulation, from Physical Agents for the Physical Therapist Assistant, FA Davis Company, 1996.
- Hooper PD: Physical Modalities-A Primer for Chiropractic, Williams & Wilkins, 1996
- Kenna KM: Pain Management with Electrical Stimulation, from Physical Agents for the Physical Therapist Assistant, FA Davis Company, 1996.
- Knight KL and Draper DO: Electrotherapy from Therapeutic Modalities: The Art and Science, Lippincott Williams & Wilkins, a Wolters Kluwer business, 2008.
- Mehreteab TA, Weisberg J and Nelson A: Electrotherapy from Physical Agents: A Comprehensive Text for Physical Therapists, Appleton & Lange, 1994.
- Mullin D and Gardner ER: Physiologic Basis of Electrical Stimulation, from Physical Agents for the Physical Therapist Assistant, FA Davis Company, 1996.
- Prentice W: Therapeutic Modalities: For Sports Medicine and Athletic Training, Mc Graw Hill Companies, 2008.
- Shapiro s: Electrical Currents from Rehabilitation: From Research to Practice, Elsevier, 2008.
- Sparrow KJ: Electrotherapeutic Modalities: Electrotherapy and Iontophoresis, from Modalities for Therapeutic Intervention (Contemporary Perspectives in Rehabilitation), F.A. Davis Company, 2005.
- 12. Starkey C: Electrical Agents, from Therapeutic Modalities, FA Davis Company, 1999.
- Stillwell GK: Electrotherapy from Krusen's Handbook of Physical Medicine and Rehabilitation, W.B. Saunders Company, 1982.

# APPENDIX PROTOCOL REVISIONS LOG

| VERSION | DATE | SIGNIFICANT REVISIONS |
|---|---|---|
| V1.0 | 6/25/2020 | Initial Release |
| V2.0 | 9/8/2021 | Expand to include extremities, strength measurements, investigators |